CLINICAL TRIAL: NCT02337361
Title: Preparing a Computerized Tool for Preventing Prenatal Drinking for a Larger Trial
Brief Title: Computerized Tool for Preventing Prenatal Drinking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Institute, California (Other)
Collaborators: Sonoma County Department of Health Services (Unknown); La Clínica de La Raza Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R34AA022697 (NIH)
Record Dates: First submitted 2014-10-21; First posted 2015-01-13 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2019-01

CONDITIONS: Foetal Exposure During Pregnancy
Keywords: risky alcohol use; pregnancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- e-SBI (Experimental): Single session, Electronic SBI for risky alcohol use
  Interventions: Behavioral: Electronic SBI
- Control (No Intervention): Treatment as usual with only assessment

INTERVENTIONS:
Behavioral: Electronic SBI — Bilingual (English and Spanish) e-SBI with four key components:
  1) Beverage-specific drink size assessment; 2) Individualized feedback on the woman's drink sizes and on discrepancies between her drink size and the standard size for each beverage; 3) A personalized plan for reducing consumption which includes goal setting; and 4) an analysis of high risk situations for drinking alcohol, and suggested coping strategies.
  Arms: e-SBI

SUMMARY:
An innovative, self-administered computerized screening and brief intervention (SBI) for drinking during pregnancy will be adapted for use with non-pregnant childbearing age women and its efficacy will be tested in a small trial. Study findings will inform a larger randomized control trial for a primary prevention tool with the potential for broad health impact.

DETAILED DESCRIPTION:
This study evaluates a recently piloted, self-administered, computerized tool for reducing prenatal drinking that added novel components of drink size assessment and drink size feedback to traditional screening and brief intervention (SBI). The bilingual (English and Spanish) electronic SBI or "e-SBI" will be adapted for use with non-pregnant women and a small trial of its efficacy will be conducted in two public health clinics. The effects of drink size assessment by itself and of depression as a modifier of e-SBI efficacy will also be studied. Study findings will help design a larger trial of e-SBI's efficacy for reducing prenatal alcohol use.

An experimental design will be used for the proposed small trial. Two hundred women, who have not been pregnant in the past year and report alcohol at risky levels will be randomly assigned to e-SBI or usual care. Participants will complete baseline, 3-month and 6-month follow-up assessments. These assessments will examine drinking and pregnancy as well as possible negative outcomes, such as increased drug use associated with the e-SBI. To address methodological limitations in prior research, the study design incorporates drink size assessment to better measure drinking outcomes, minimizes assessment reactivity for controls at baseline, and includes a booster e-SBI at the 3-month follow up. This allows for the examination of whether drink size assessment reduces drinking by itself and if its effects are equivalent to that of the full e-SBI. With these design innovations, the study is expected to provide information that can be more rigorously assessed in a subsequent multi-arm trial. Because it sets the stage for a Phase II trial of e-SBI efficacy for reducing prenatal alcohol use, our proposed study is of significance for improved maternal and child health. Findings will also impact the larger intervention literature on cost-effective strategies to reduce alcohol-related harm.

ELIGIBILITY:
Inclusion Criteria:

* not pregnant in the last 6 months, drank alcohol in the past year, alcohol consumption was at risky levels,

Exclusion Criteria:

* not fluent in english or spanish,

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 185 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhabika Nayak, Ph.D., Principal Investigator — Public Health Institute
Locations (2):
- United States (2):
  - La Clinica Women Infants and Children Program Site, Oakland, California
  - Sonoma County Department of Health Services, Santa Rosa, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nayak MB, Kaskutas LA, Mericle AA. Randomized Trial of an Innovative Electronic Screening and Brief Intervention for Reducing Drinking Among Women of Childbearing Age. J Addict Med. 2019 Nov/Dec;13(6):450-459. doi: 10.1097/ADM.0000000000000518. PMID 30882553

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant was assigned to control group but did not complete baseline assessment
Groups:
- e-SBI: Single session, Electronic Screening and Brief Intervention (SBI) for risky alcohol use
  Electronic SBI: Bilingual (English and Spanish) e-SBI with four key components:
  1) Beverage-specific drink size assessment; 2) Individualized feedback on the woman's drink sizes and on discrepancies between her drink size and the standard size for each beverage; 3) A personalized plan for reducing consumption which includes goal setting; and 4) an analysis of high risk situations for drinking alcohol, and suggested coping strategies.
Period: Baseline Assessment
Arm/Group | e-SBI | Control
Started | 99 | 86
Completed | 99 | 86
Not Completed | 0 | 0
Period: 3-month Follow-up
Arm/Group | e-SBI | Control
Started | 99 | 86
Completed | 80 | 72
Not Completed | 19 | 14
Not completed — Lost to Follow-up | 19 | 14
Period: 6-month Follow-up
Arm/Group | e-SBI | Control
Started | 80 | 72
Completed | 78 | 68
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- e-SBI: Single session, Electronic SBI for risky alcohol use
  Electronic SBI: Bilingual (English and Spanish) e-SBI with four key components:
  1) Beverage-specific drink size assessment; 2) Individualized feedback on the woman's drink sizes and on discrepancies between her drink size and the standard size for each beverage; 3) A personalized plan for reducing consumption which includes goal setting; and 4) an analysis of high risk situations for drinking alcohol, and suggested coping strategies.
- Total: Total of all reporting groups
Arm/Group | e-SBI | Control | Total
Number analyzed (Participants) | 99 | 86 | 185
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 99 | 86 | 185
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 86 | 185
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 72 | 66 | 138
  Not Hispanic or Latino | 27 | 20 | 47
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 99 | 86 | 185
Risky alcohol use [Count of Participants; unit: Participants] — Risky alcohol use is defined as drinking 8 or more drinks in a week or 3 or more drinks in a day.
  to be enrolled in the trials as risky drinkers, participants had to meet these criteria for risky alcohol use.
  Participants | 99 | 86 | 185

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Risky Alcohol Use
Description: Risky alcohol use is defined as drinking 8 or more drinks in a week or 3 or more drinks in a day.
  Risky alcohol use is measured by frequency of any alcohol use, number of usual and maximum drinks in a drinking day, and frequency of drinking 3 or more drinks containing alcohol
Time Frame: baseline, 3 months, 6 months
Population: 3 and 6 month numbers for each arm (study condition) reflect participant attrition over time
Measure: Count of Participants; unit: Participants
Arm/Group | e-SBI | Control
Number analyzed (Participants) | 99 | 86
Participants
  baseline | 99 | 86
  3 month: number analyzed (Participants) | 80 | 72
  3 month | 60 | 48
  6 month: number analyzed (Participants) | 78 | 68
  6 month | 45 | 41
Statistical Analysis 1: Comparison: Control; Test type: Other; Generalized estimating equations (GEE)(Diggle et al. 2002) tested e-SBI efficacy, controlling for demographic differences between study condition and study sites. GEE models estimate population average or marginal models and account for within-subject nonindependence (clustering) of observations across multiple waves of data collection and use all available data in model estimation
Statistical Analysis 2: Comparison: Control; Test type: Other; Generalized estimating equations tested e-SBI efficacy, controlling for demographic differences between study condition and study sites. GEE models estimate population average or marginal models and account for within-subject nonindependence (clustering) of observations across multiple waves of data collection and use all available data in model estimation

2. Primary Outcome: Number of Participants Reporting Weekly Alcohol Use
Description: weekly alcohol use is defined as at least drinking once a week or more often
Time Frame: baseline, 3 month, 6 month
Population: 3 and 6 month numbers for each arm (study condition) reflect participant attrition over time
Measure: Count of Participants; unit: Participants
Arm/Group | e-SBI | Control
Number analyzed (Participants) | 99 | 86
Participants
  Baseline | 22 | 14
  3 month: number analyzed (Participants) | 80 | 72
  3 month | 17 | 16
  6 month: number analyzed (Participants) | 78 | 68
  6 month | 9 | 16
Statistical Analysis 1: Comparison: Control; Test type: Other; p < .01, t-test, 2 sided; Odds Ratio (OR) = 0.22, Standard Error of Mean 0.12 — the e-SBI group was at reduced odds relative to the control group to report weekly or more frequent drinking at 6 month follow-up; Generalized estimating equations (GEE) tested e-SBI efficacy, controlling for demographic differences between study condition and study sites. GEE models estimate population average or marginal models and account for within-subject nonindependence (clustering) of observations across multiple waves of data collection and use all available data in model estimation

3. Primary Outcome: Number of Participants Reporting Heavy Alcohol Use
Description: heavy alcohol use is defined as self-reported maximum number of drinks in a day of 5 or more drinks
Time Frame: baseline, 3 month, 6 month
Population: Numbers at 3 and 6 month reflect participant attrition
Measure: Count of Participants; unit: Participants
Arm/Group | e-SBI | Control
Number analyzed (Participants) | 99 | 86
Participants
  Baseline | 19 | 16
  3 month: number analyzed (Participants) | 80 | 72
  3 month | 14 | 18
  6 month: number analyzed (Participants) | 78 | 68
  6 month | 7 | 16
Statistical Analysis 1: Comparison: Control; Test type: Other; p < .05, t-test, 2 sided; Odds Ratio (OR) = 0.23, Standard Error of Mean 0.14 — the e-SBI group was at reduced odds relative to the control group to report drinking a maximum quantity of 5 or more drinks in a day at 6 month follow-up

4. Secondary Outcome: Number of Participants Reporting Any Tobacco Use
Description: Any Tobacco use is measured as any use in the past 3 months of any smoking or chewing tobacco, including cigarettes
Time Frame: baseline , 3 months, 6 months
Population: numbers at follow up reflect participant attrition over time
Measure: Count of Participants; unit: Participants
Arm/Group | e-SBI | Control
Number analyzed (Participants) | 99 | 86
Participants
  Baseline | 20 | 16
  3 month: number analyzed (Participants) | 80 | 72
  3 month | 12 | 11
  6 month: number analyzed (Participants) | 78 | 68
  6 month | 9 | 13
Statistical Analysis 1: Comparison: Control; Test type: Other; p < .10, t-test, 2 sided; Odds Ratio (OR) = 0.51, Standard Error of Mean 0.20 — the e-SBI group was at reduced odds relative to the control group to report any tobacco use at 6 month follow-up; [other analysis details as in outcome 2, analysis 1]

5. Secondary Outcome: Number of Participants Reporting Frequent Sugar Sweetened Beverage Use
Description: Frequent Sugar sweetened beverage use is defined as at least weekly consumption of sugar sweetened beverages
Time Frame: baseline, 3 months, 6 months
Population: numbers at 3 and 6 month reflect participant attrition over time
Measure: Count of Participants; unit: Participants
Arm/Group | e-SBI | Control
Number analyzed (Participants) | 99 | 86
Participants
  Baseline | 65 | 58
  3 month: number analyzed (Participants) | 80 | 72
  3 month | 55 | 46
  6 month: number analyzed (Participants) | 78 | 68
  6 month | 41 | 33
Statistical Analysis 1: Comparison: Control; Test type: Other; p < .01, t-test, 2 sided; Odds Ratio (OR) = 0.26, Standard Error of Mean 0.15 — the e-SBI group was at reduced odds relative to the control group to report significant depression at 6 month follow-up

6. Secondary Outcome: Number of Participants Reporting Significant Depression
Description: Significant depression is measured as scoring above the cutoff of 6 on the total score on the 9 item Physician's health questionnaire (PHQ-9).
  The 9-item Patient Health Questionnaire (PHQ-9) is a self-report measure of depression symptoms in the past two weeks. Scores can range from 0 to 27, with a score of 6 or more indicating significant depression symptoms in samples of childbearing age women.
Time Frame: baseline, 3 months, 6 months
Population: numbers at 3 and 6 month reflect participant attrition over time
Measure: Count of Participants; unit: Participants
Groups:
- Control: Treatment as usual, No intervention
Arm/Group | e-SBI | Control
Number analyzed (Participants) | 99 | 86
Participants
  Baseline | 22 | 11
  3 month: number analyzed (Participants) | 80 | 72
  3 month | 16 | 12
  6 month: number analyzed (Participants) | 78 | 68
  6 month | 8 | 11
Statistical Analysis 1: Comparison: Control; Test type: Other; Generalized estimating equations (GEE) tested DrinkWise's effects on changes in depression over time controlling for demographic differences between study condition and study sites

7. Secondary Outcome: Number of Participants Reporting Any Drug Use
Description: Any drug use is defined as use of any substances, e.g., marijuana, stimulants, etc other than tobacco, in the past 3 months
Time Frame: baseline, 3 month, 6 month
Population: numbers at 3 and 6 month reflect participant attrition over time
Measure: Count of Participants; unit: Participants
Arm/Group | e-SBI | Control
Number analyzed (Participants) | 99 | 86
Participants
  Baseline | 12 | 10
  3 month: number analyzed (Participants) | 80 | 72
  3 month | 8 | 6
  6 month: number analyzed (Participants) | 78 | 68
  6 month | 9 | 5

ADVERSE EVENTS:
Time Frame: 18 months, 6 months per participation, overall time frame includes screening for eligibility until the completion of the last (6-month follow-up) for the participants enrolled into the study last
Description: The trial did not involve drugs or biologics, devices, or invasive procedures and involved a behavioral intervention with no known risks to participants.
  Drinking and mental health behaviors included in outcomes were assessed at each follow up. But no adverse events were observed any time in the study.
Arm/Group | e-SBI | Control
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/86
Other Adverse Events (participants affected / at risk) | 0/99 | 0/86

LIMITATIONS AND CAVEATS:
Participants in the e-SBI group were re-administered the brief intervention at 3-month follow-up if they reported any alcohol use at that follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2015-06-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT02337361/SAP_000.pdf
  • Study Protocol (2015-06-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT02337361/Prot_001.pdf